CLINICAL TRIAL: NCT03673488
Title: Prospective Study to Evaluate Use of TephaFLEX™ Sling Implanted Via a Retropubic Mid-urethral Sling Procedure for Treatment of Women With Stress Urinary Incontinence
Brief Title: To Evaluate the Use of Bioresorbable Tephaflex™ Sling for Stress Urinary Incontinence
Acronym: Tephaflex
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Pelvic Floor Research Foundation of South Africa (Other)
Collaborators: University of Cape Town (Other)
Responsible Party: Sponsor
Other Study IDs: URO001
Record Dates: First submitted 2018-09-03; First posted 2018-09-17 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Stress Urinary Incontinence
Keywords: Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TephaFlex™ mid-urethral sling for SUI: P4HB material ( TephaFlex ™) will be implanted in 25 women with confirmed Stress Urinary Incontinence (SUI).
  Interventions: Device: TephaFlex™ mid-urethral sling

INTERVENTIONS:
Device: TephaFlex™ mid-urethral sling — The sling is made from P4HB material. It is placed in a similar technique to standard retropubic sling procedures, but will resorb over 18-24 months post surgery.
  Other Names: P4HB mid-urethral bioresorbable sling

SUMMARY:
Urinary incontinence (UI) is a major public health issue affecting up to 25-50% of all women and has a detrimental impact on patient quality of life. Stress urinary incontinence (SUI) is the most common form of urinary incontinence and is defined as the leakage of urine, which occurs during physical activity of exertion or on sneezing or coughing. It has been reported that the prevalence of SUI is 25 to 45% of the female population. If pelvic floor exercises are not effective, mid-urethral slings (MUS) are widely used as a first-line surgical treatment. Subjective and objective cure rates of 91% and 85% respectively have been reported for retropubic midurethral slings.

Midurethral slings are commonly made of polypropylene (PP). Although the polypropylene products are effective and have relatively low rates of adverse events, the adverse events that do occur, like exposure and pain, have been related to the fact that a permanent synthetic mesh is implanted. Mesh-related complications are difficult to manage and may even involve partial or complete removal of the implant.

Clinically, there is a need to investigate whether mid-urethral sling surgery can be performed with a non-permanent mesh made from a resorbable biomaterial, as an alternative for PP. Non-permanent meshes may be associated with fewer complications and better quality of life. However, before non-permanent and permanent mesh procedures can be compared, there is a need to first establish the feasibility of using a mesh in a mid-urethral sling procedure.

The investigators hypothesize that a retropubic mid-urethral sling procedure to treat stress urinary incontinence, can be successfully performed using an implant made of poly-4-hydroxybutyrate (P4HB).

DETAILED DESCRIPTION:
The overall objective of this study is to determine the preliminary safety and efficacy of resorbable TephaFLEX sling implanted via a retropubic procedure to treat SUI.

Prospective, observational single-center study with a follow-up of 24 months post-surgery. Up to 25 patients will be recruited at Groote Schuur Hospital Urogynecology Out-Patient Department. Eligible patients will receive a retropubic surgical producedure where a TephaFLEX sling, composed of the resorbable material P4HB, is placed. After the surgical procedure, follow-up visits are scheduled at 4-6 weeks, 3 months (+/- 2 weeks), 6 months (+/- 2 weeks), 12 months (+/- 1 month), and 24 months (+/- 1 month) post-procedure. TephaFLEX sling, manufactured by Tepha, Inc., will be implanted via a retropubic mid-urethral sling procedure for treatment of women with stress urinary incontinence. The product is supplied as a sterile, single-use device. One device will be utilized per patient. TephaFLEX sling, developed specifically for treatment of stress urinary incontinence, is a single layer, bioresorbable, mesh made from poly-4-hydroxybutyrate (P4HB) monofilament fiber. The mesh is constructed as a 11mm x 60cm tape with an open pore structure, and is enclosed in a polyethylene sleeve to ease insertion. The mesh was designed specifically to provide strength over the three-month critical wound healing period in soft tissue repair and reinforcement, and to encourage the proliferation of healthy tissue at the repair site. The product undergoes a gradual loss of strength after implantation and is essentially resorbed by 18 - 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Be female, = 18 years of age
2. Female symptomatic (moderate or severe) SUI resulting from urethral hypermobility and/or intrinsic sphincter deficiency (ISD).
3. Patients who have planned to undergo surgical correction of symptomatic SUI after consultation with their physician about the risks and benefits of such a procedure, and a determination by the physician that surgical treatment is the most appropriate treatment option for the patient.
4. Understand and be willing to follow all aspects of the study protocol and have signed and dated the EC-approved Informed Consent prior to any study-related procedures being performed

Exclusion Criteria:

1. Subjects who have mixed or urge incontinence
2. Subjects who have stage 2 or more genital prolapse, according to the ICS classification
3. Subjects with previous surgery for SUI
4. Subjects who undergo concomitant surgical procedures
5. Subjects who are pregnant or want to become pregnant in the next 24 months
6. Subjects who are not capable of giving informed consent
7. Subjects with a BMI = 35 kg/m2
8. Subjects diagnosed with a current urinary tract infection or chronic urinary tract infections (defined as 4 or more UTI in the last year)
9. Subjects with known sensitivity to tetracycline or kanamycin

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population are eligible women, older than 18 years of age, with demonstrable stress urinary incontinence who present to the Out-Patient Department for Urogynaecology at Groote Schuur Hospital in Cape Town South Africa. Groote Schuur Hospital is a tertiary academic hospital and serves the city of Cape Town and surrounds.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2018-06-22 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Device safety will be established by measuring the incidence of treatment-emergent adverse events. | 2 years
  The retropubic mid-urethral sling procedure using UroFLEX sling is considered to be safe at 6 months after implantation if the number of serious adverse events comply with safety standards as defined by the safety criteria outlined below and analyzed using sequential analysis. The device will be considered safe at A) a maximum of 3 of the first 5 patients experience a device or procedure-related SAE (60%); B) a maximum of 5 of the first 10 patients experience a device or procedure-related SAE (50%); C) a maximum of 7 of the first 20 patients experience a device or procedure-related SAE (35%); D) a maximum of 8 of the first 25 patients experience a device or procedure-related SAE (32%).

SECONDARY OUTCOMES:
Objective cure measurement using Cough Stress Test | Measured at enrolment, 4-6 weeks, 3, 6, 12 and 24 months post procedure (2 years total)
  Preliminary effectiveness will be assessed by measuring the number of patients that exhibit objective cure based on Cough Stress Test
Subjective cure with PGI-I questionnaire Patient Global Impression of Improvement | Administered at 4-6 weeks, 3, 6, 12 and 24 months post procedure (2 years total)
  Number of patients that exhibit subjective cure based on PGI-I questionnaire.
Subjective cure with Sandvik scores (Incontinence severity index) | Administered at 4-6 weeks, 3, 6, 12 and 24 months post procedure (2 years in total)
  Number of patients showing subjective cure on Sandvik scores questionnaire
Subjective cure with PISQ-IR- Sexual Function for Women with Pelvic Organ Prolapse, Urinary Incontinence and / or Fecal Incontinence questionnaire | Administered at 4-6 weeks, 3, 6,12,24 months post procedure (2 years in total)
  Number of patients showing subjective cure using the PISQ-IR questionairre as measurement
Subjective cure with Urogenital Distress Inventory (UDI-6) | Administered at 4-6 weeks, 3,6,12 and 24 months post procedure ( 2 years in total)
  Number of patients showing subjective cure using the UDI-6

CONTACTS AND LOCATIONS:
Overall Officials: Jan-Paul Roovers, MD, Study Chair — Pelvic Floor Research Foundation of South Africa
Locations (1):
- Groote Schuur Academic Hospital, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: No